CLINICAL TRIAL: NCT01996527
Title: Early Detection of Glioma Treatment Response Using MRI-Based Biomarkers
Brief Title: 3T MRI Biomarkers of Glioma Treatment Response
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Thomas Yankeelov, Professor of Radiology and Radiological Sciences, Director of Cancer Imaging Research, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VICC NEU 1268; NCI-2013-02195 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA068485 (NIH)
Record Dates: First submitted 2013-11-15; First posted 2013-11-27 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Diffusion Magnetic Resonance Imaging; Dynamic Contrast Enhanced Magnetic Resonance Imaging; Perfusion Magnetic Resonance Imaging; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3-Tesla magnetic resonance imaging (Experimental): Patients undergo 3-Tesla magnetic resonance imaging to measure tumor protein content (using CEST-MRI), cellularity (using DW-MRI), and blood flow (using DCE-MRI and DSC-MRI with IV administration of gadolinium-containing contrast agent) no more than 2 weeks before, and 2 and 4 weeks after, the initiation of treatment.
  Interventions: Device: 3-Tesla magnetic resonance imaging; Device: CEST-MRI; Device: DW-MRI; Device: DCE-MRI; Device: DSC-MRI; Drug: IV administration of gadolinium-containing contrast agent

INTERVENTIONS:
Device: 3-Tesla magnetic resonance imaging — 3-Tesla MRI is a multiparametric imaging exam that includes MR pulse sequences for CEST-MRI, DW-MRI, DCE-MRI, and DSC-MRI
  Other Names: 3-Tesla MRI; 3T MRI
Device: CEST-MRI — Undergo CEST-MRI
  Other Names: chemical exchange saturation transfer MRI
Device: DW-MRI — Undergo DWI-MRI
  Other Names: diffusion-weighted MRI
Device: DCE-MRI — Undergo DCE-MRI
  Other Names: dynamic contrast-enhanced MRI
Device: DSC-MRI — Undergo DSC-MRI
  Other Names: dynamic susceptibility contrast MRI
Drug: IV administration of gadolinium-containing contrast agent — Gadolinium-containing paramagnetic contrast agent (Magnevist®; Berlex Lab, Wayne, New Jersey) in delivered via intravenous (IV) infusion to achieve DCE and DSC contrast
  Other Names: Magnevist®; gadopentetate dimeglumine

SUMMARY:
This pilot clinical trial studies advanced magnetic resonance imaging (MRI) techniques in measuring treatment response in patients with high-grade glioma. New diagnostic procedures, such as advanced MRI techniques at 3 Tesla, may be more effective than standard MRI in measuring treatment response in patients receiving treatment for high-grade gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To correlate treatment-induced changes in quantitative MRI-based biomarkers-specifically, those sensitive to tumor protein content (amide proton transfer asymmetry [APTasym] from chemical exchange saturation transfer [CEST]), cellularity (apparent diffusion coefficient [ADC] from diffusion-weighted imaging [DWI]), and blood flow (volume transfer constant [K^trans] from dynamic contrast-enhanced [DCE]; cerebral blood flow [CBF] from dynamic susceptibility contrast [DSC])-with treatment-induced changes in tumor size, measured via standard anatomic MRI.

II. To correlate treatment-induced changes in the above quantitative MRI endpoints with patient progression-free survival (PFS).

OUTLINE:

Patients undergo measurement of tumor protein content using CEST-MRI, cellularity using DWI-MRI, and blood flow using DCE-MRI and DSC-MRI within 2 weeks of treatment and at 2 and 4 weeks after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign an institutional review board (IRB)-approved informed consent document
* Patients must have been diagnosed with high-grade glioma:

  * World Health Organization (WHO) grade III: anaplastic astrocytoma, oligodendroglioma, ependymoma, or oligoastrocytoma; OR
  * WHO grade IV: glioblastoma multiforme; or neuroepithelial tumors of uncertain origin (polar spongioblastoma, astroblastoma, or gliomatosis cerebri)
* As measured by conventional high spatial resolution MRI, the minimum diameter of the primary lesion (short axis) should be at least 5 mm
* Patients must be scheduled to receive: 1) standard chemotherapy with/without radiation therapy; OR 2) single-agent bevacizumab (Avastin)

Exclusion Criteria:

* Patients with low-grade (WHO grade I or II) glioma
* Patients with metastatic disease
* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who have any type of ferromagnetic bioimplant that could potentially be displaced
* Patients who have cerebral aneurysm clips
* Patients who may have shrapnel imbedded in their bodies (such as from war wounds), metal workers and machinists (potential for metallic fragments in or near the eyes)
* Patients with inadequate renal function (creatinine >= 1.5 times upper limit of normal) or acute or chronic renal insufficiency (glomerular filtration rate < 20 ml/min)
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential
* Patients who exhibit noticeable anxiety and/or claustrophobia or who exhibit severe vertigo when they are moved into the magnet bore
* Patients incapable of giving informed written consent, for the following reasons:

  * Inability to adhere to the experimental protocols for any reason
  * Inability to communicate with the research team
  * Limited ability to give informed consent due to mental disability, altered mental status, confusion, cognitive impairment, or psychiatric disorders

    * Patients scoring 14.5 or lower on the University of California at San Diego (UCSD) Brief Assessment of Consent Capacity (UBACC) Capacity to Consent Questionnaire will be excluded
  * Prisoners or other individuals deemed to be susceptible to coercion
* For patients who have undergone surgical resection prior to joining the study, in whom baseline magnetic resonance (MR) images exhibit enough signal degradation (due to susceptibility artifact in the region of the surgical bed) such that the data are uninterpretable will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11-23 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Best Response | On-treatment date to date of disease progression (up to 12 weeks)
  Number of patients in each response category, per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, summarized as follows for target lesion criteria: complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter (LD) of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | On-study date to lesser of date of progression or date of death from any cause (assessed at 6 months)
  Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring. Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters (LD) of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.

OTHER OUTCOMES:
Changes in quantitative MRI-based biomarkers sensitive to tumor protein content | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Amide proton transfer asymmetry (APTasym, %) from CEST
Changes in quantitative MRI-based biomarkers sensitive to tumor cellularity and vascularity | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Apparent diffusion coefficient (ADC, mm2/s) from DW-MRI
  2. Tissue diffusion coefficient (Dt, mm2/s) from DW-MRI
  3. Pseudo-diffusion coefficient (Dp, mm2/s) from DW-MRI
Changes in quantitative MRI-based biomarkers sensitive to tumor perfusion and hemodynamics | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Volume transfer constant (Ktrans, 1/min) from DCE-MRI
Changes in quantitative MRI-based biomarkers sensitive to tumor perfusion and hemodynamics | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Perfusion fraction (fp, %) from DW-MRI
  2. Extravascular extracellular volume fraction (ve, %) from DCE-MRI
  3. Plasma volume fraction (vp, %) from DCE-MRI
  4. Cerebral blood volume (CBV, %) from DSC-MRI
Changes in quantitative MRI-based biomarkers sensitive to tumor perfusion and hemodynamics | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Cerebral blood flow (CBF, ml/min/100 g) from DSC-MRI
Changes in quantitative MRI-based biomarkers sensitive to tumor perfusion and hemodynamics | Baseline to within 4 weeks after on-treatment date
  Evaluation of the following biological imaging metrics:
  1. Mean transit time (MTT, s) from DSC-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Chad Quarles, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct